CLINICAL TRIAL: NCT02921152
Title: Bone Marrow Micrometastases in Patients With Early Stage Breast Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Acibadem University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ATADEK 2015/11
Record Dates: First submitted 2016-05-17; First posted 2016-10-03 (Estimated); Last update posted 2016-10-03 (Estimated); Status verified 2016-08

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- all (Other): All patients with early breast cancer
  Interventions: Procedure: bone marrow aspiration /trephine biopsy

INTERVENTIONS:
Procedure: bone marrow aspiration /trephine biopsy

SUMMARY:
Operable early stage breast cancer patients staged according to NCCN guidelines are subjected to bone marrow aspiration/trephine biopsy at the time of the definitive operation under general anesthesia. The specimen will be fixated in neutral tamponaded formalin and the sections will be examined by H&E and cytokeratin immunohistochemically. If disseminated tumor cells are identified ER (estrogen receptor), PR (progesterone receptor), HER2/neu will be studied. Disseminated tumor cells will be recorded quantitively and semiquantitatively. Results of the pilot study will be evaluated as observational study.

ELIGIBILITY:
Inclusion criteria:

1. Patients over 18 years old and who have given informed consent to enter the study.
2. ASA I-II patients
3. Patients who have not been diagnosed as breast cancer or received any type of treatment regarding breast cancer before the time of study
4. Patients who are appropriate for bone marrow biopsy
5. Menopausal status is not relevant.

Exclusion criteria:

1. Active collagen tissue disorders
2. Patients who are diagnosed having breast cancer and received any type of treatment regarding breast cancer before the time of study
3. Pregnancy
4. Patients with bleeding disorders, who are receiving antiaggregant or anticoagulant medication.
5. Patients who refused to enter the study protocol and refused to give informed consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2016-04; Primary Completion 2018-04 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Rate of bone marrow metastases in early stage breast cancer | up to 5 years
  Number of patients with bone marrow metastases/ total number of enrolled patients
Rate of sentinel lymph node metastases in early stage breast cancer | up to 5 years
Rate of sentinel lymph node metastases in patients with bone marrow metastasis operated for early stage breast cancer | up to 5 years
Incidence of bone marrow metastasis in HER-2 positive early stage breast cancer | up to 5 years
Incidence of bone marrow metastases in triple negative early stage breast cancer | up to 5 years

SECONDARY OUTCOMES:
Incidence of axillary recurrence in patients with negative sentinel lymph node biopsy | Up to 10 years
Overall survival | up to 10 years

OTHER OUTCOMES:
Disease free survival | up to 10 years

CONTACTS AND LOCATIONS:
Locations (1):
- Acibadem University School of Medicine, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided